CLINICAL TRIAL: NCT03100162
Title: Effect of Oral Supplementation With Probiotics on Cardiometabolic Risk Factors, Microflora and Intestinal Epithelial Permeability, Mineral Content and Lifestyle in Obese Women With Postmenopausal Metabolic Syndrome: Double-blind, Randomized Clinical Trial.
Brief Title: Effect of Oral Supplementation With Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: German Institute of Human Nutrition Potsdam-Rehbruecke (DIfE) (Unknown); Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Pawel Bogdanski, Professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 871/15
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: probiotics; metabolic syndrome; obesity; microbiome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Individuals receive a placebo daily, for 3 months.
  Interventions: Dietary Supplement: Placebo
- Probiotic 2g (Active Comparator): Individuals receive 2 g of probiotic daily, for 3 months.
  Interventions: Dietary Supplement: Probiotic
- Probiotic 4g (Active Comparator): Individuals receive 4 g of probiotic daily, for 3 months.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic 2g; Probiotic 4g
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Effect of oral supplementation with probiotics on cardiometabolic risk factors, microflora and intestinal epithelial permeability, mineral content and lifestyle in obese women with postmenopausal metabolic syndrome: double-blind, randomized clinical trial.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether oral probiotic supplementation affects cardiometabolic risk, intestinal epithelial permeability, metabolic activity and intestinal flora composition, mineral content, and lifestyle in obese women with metabolic syndrome.

Probiotics are a group of non-pathogenic microbes that bring health benefits to the host. Their use enables the variety and proper functioning of intestinal microflora. The use of probiotics increases the amount of bifidobacteria and lactobacilli, what directly affects the reduction of endotoxemia by sealing the intestinal wall, as well as the improvement of fat, carbohydrate and insulin metabolism.

The project is due to evaluate the effect of supplementation with selected probiotics in patients with metabolic syndrome on:

* lipid metabolism- total cholesterol, HDL and LDL cholesterol and triglycerides,
* blood glucose concentration,
* blood pressure values,
* anthropometric parameters,
* quality of life,
* the contentl of minerals,

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) equal to or greater than 30 kg/m2
* age 45 to 70 years
* stable body weight (< 3 kg self-reported change during the previous three months)
* written informed consent to participate in the study,
* > = 1 year after the last menstrual period;
* abdominal obesity - waist circumference> 80 cm;
* body fat content measured by bio-impedance ≥ 33%;

Exclusion Criteria:

* secondary obesity or secondary hypertension
* diabetes type I
* gastrointestinal disease;
* dyslipidaemia, type 2 diabetes, hypertension requiring the implementation of pharmacological treatment in the last 3 months prior to observation or follow-up;
* a history of use of any dietary supplements within the one month prior to the study
* taking antibiotics within 1 month before starting the study;
* Clinically relevant acute or chronic inflammatory disease in the respiratory, gastrointestinal or genitourinary system or in the mouth, throat, paranasal sinuses and / or connective tissue disease, arthritis;
* simultaneous participation in a study that affects weight change or use of diet / medication / nutritional behaviors affecting body weight changes;
* consumption of pre- and probiotic-enriched products (for at least 3 weeks prior to the first screening visit) and products with high fiber content or large amounts of fermented foods (> 400g / day);
* hormone replacement therapy;
* a history of infection in the month prior to the study
* nicotine, drug or alcohol abuse
* vegetarian diet;
* or other condition that, in the opinion of the investigators, would make participation not in the best interest of the patient or could prevent, limit, or confound the study results

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2016-02-27 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with decreased cardiometabolic risk | At the baseline and after 3 months of treatment
  Cardiometabolic risk will be estimated at baseline and after 3 months of treatment using the SCORE scale. SCORE scale summarize 5 risk factors (sex, age, systolic blood pressure, total cholesterol and smoking). The number of patients with decreased cardiometabolic risk will be measured.

SECONDARY OUTCOMES:
blood pressure | At the baseline and following 3 months of treatment
Body mass index | At the baseline and following 3 months of treatment
waist circumference | At the baseline and following 3 months of treatment
serum lipids | At the baseline and following 3 months of treatment
Total antioxidant status (TAS) evaluated by colorimetric method with Tas Randox kit | At the baseline and following 3 months of treatment
insulin estimated by immunoassay (DIAsource immunoassays) | At the baseline and following 3 months of treatment
interleukin-6 measured by an enzyme-linked immunosorbent assay (R&D Quantikine® Human Il-6 kit) | At the baseline and following 3 months of treatment
Total body fat content | At the baseline and following 3 months of treatment
  Total body fat content will be measured at baseline and after 3 months of treatment using electrical bioimpedance
Measurement of mineral content in hair | At the baseline and following 3 months of treatment
  The content of iron, magnezium, calcium, selenium, copper and lead in patients' hair at baseline and after 3 months of treatment will be estimated using atomic absorption spectrometry.
Fecal examination (Kalprotektyna, Alfa1 - antytrypsyna ) | At the baseline and following 3 months of treatment
Quality of life | At the baseline and following 3 months of treatment
  "The World Health Organization Quality of Life (WHOQOL) - BREF"

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Bogdanski, MD PhD, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Department of Education and Obesity Treatment and Metabolic Disorders, Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided